CLINICAL TRIAL: NCT05928741
Title: Short-term Effects of Fruit Juice Enriched With Vitamin D3, n-3 Fatty Acids, and Probiotics on Subjective Appetite, Energy Intake, and Glycemic Responses, in Healthy Adults
Brief Title: Short-term Effects of Juice Consumption With Biofunctional Compounds and Probiotics on Subjective Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: HRBD 73/04.10.2022
Record Dates: First submitted 2023-06-24; First posted 2023-07-03 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Subjective Appetite
Keywords: subjective appetite; feeding behavior; glycemic responses; enriched juice; probiotics; vitamin D3; n-3 fatty acids
MeSH Terms: conditions — Feeding Behavior | interventions — Cholecalciferol; Fatty Acids, Omega-3; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind (participant, investigator, outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orange juice with vitamin D3, n-3 fatty acids, and probiotics as preload (Experimental): Twenty-three healthy adults with normal weight and twenty-three healthy adults with overweight consumed a standardized breakfast after a 12-hour fast. Two hours later they were given 50 g of available carbohydrates from the two preloads (enriched orange juice or control orange juice) in a random order, and 3 hours after the preload they were offered an ad libitum lunch. Foods were weighed at the time of serving and any leftovers were weighed again after lunch to determine the amount of food consumed. There was a washout period of at least one week between the two visits. Fingertip capillary blood glucose samples were collected at baseline and at several time points after food intake. Visual analog scales (VAS) of 100 mm were collected to assess subjective appetite. Blood pressure was measured at several time-points.
  Interventions: Behavioral: Orange juice with vitamin D3, n-3 fatty acids, and probiotics as preload
- Control orange juice without vitamin D3, n-3 fatty acids, and probiotics as preload (Experimental): Twenty-three healthy adults with normal weight and twenty-three healthy adults with overweight consumed a standardized breakfast after a 12-hour fast. Two hours later they were given 50 g of available carbohydrates from the two preloads (enriched orange juice or control orange juice) in a random order, and 3 hours after the preload they were offered an ad libitum lunch. Foods were weighed at the time of serving and any leftovers were weighed again after lunch to determine the amount of food consumed. There was a washout period of at least one week between the two visits. Fingertip capillary blood glucose samples were collected at baseline and at several time points after food intake. Visual analog scales (VAS) of 100 mm were collected to assess subjective appetite. Blood pressure was measured at several time-points.
  Interventions: Behavioral: Orange juice with vitamin D3, n-3 fatty acids, and probiotics as preload

INTERVENTIONS:
Behavioral: Orange juice with vitamin D3, n-3 fatty acids, and probiotics as preload — Twenty-three healthy adults with normal weight and twenty-three healthy adults with overweight consumed a standardized breakfast consisting of 2 slices of white bread and honey (350 kcal in total) after a 12-hour fast. Two hours later they were offered 347 mL of the enriched orange juice (containing 50 g available carbohydrates), and 3 hours after the preload they were offered an ad libitum lunch (chicken breast with white rice). Foods were weighed at the time of serving and any leftovers were weighed again after lunch to determine the amount of food consumed. Fingertip capillary blood glucose samples and visual analog scales (VAS) of 100 mm were collected at baseline and at 60, 120, 135, 150, 180, 210, 240, 270, 300, 330, 360, 390, and 420 minutes after breakfast consumption. Blood pressure was measured at baseline, 120, 300, and 420 minutes.

SUMMARY:
This study investigated the short-term effects of fruit juice enriched with vitamin D3, n-3 fatty acids, and probiotics on subjective appetite, energy intake, and glycemic responses, in both normal-weight and overweight, healthy adults.

DETAILED DESCRIPTION:
This study aimed to 1. Assess the subjective appetite of participants after the consumption of fruit juice (100% orange) enriched with vitamin D3, n-3 fatty acids, and probiotics compared to regular fruit juice (without any fortification), and 2. Examine the short-term effects of enriched fruit juice compared to regular fruit juice on glycemic responses and blood pressure, in both normal-weight and overweight healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Healthy Non-diabetic men and women Body mass index between 18.5 and 29.9 kg/m2

Exclusion Criteria:

* Severe chronic disease (i.e., cardiovascular diseases, diabetes mellitus, kidney or liver conditions, endocrine conditions)
* Gastrointestinal disorders
* Pregnancy
* Lactation
* Competitive sports
* Alcohol abuse
* Drug dependency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Subjective appetite rating | 7 hours
  Useful change in subjective appetite using visual analogue scales (VAS). Participants rated their hunger, desire to eat, perceived fullness, thirst, preoccupation with food, pleasure of eating the consumed test food, and thirst, after eating on a horizontal line VAS, with a line length of 100 mm and width of 3 desktop publishing points, that was black, had flat line endpoints, had an ascending numerical order of scale endpoints [i.e., "0" and "10", for example neither hungry (0 mm), full (100 mm) or have desire for food in the middle (50 mm)], and used "0" and "100" as numerical anchors below the left and right endpoints, respectively.

SECONDARY OUTCOMES:
Energy intake after preload and the next 24 hours | 24 hours
  Clinically significant difference in energy intake (ad libitum lunch) two hours after the two different preloads consumption, as well as the next 24 hours after the intervention (actual weighing of foods consumed and leftovers, and 24-hour recall).

OTHER OUTCOMES:
Capillary blood glucose responses | 7 hours
  Clinically significant change in capillary blood glucose levels between the two interventions.
Blood pressure | 7 hours
  Clinically significant change in systolic and diastolic blood pressure between the two interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Aimilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece